CLINICAL TRIAL: NCT02139033
Title: A Single-Center Evaluation of Retaine™ Ophthalmic Emulsion in the Management of Tear Film Stability and Ocular Surface Staining in Patients Diagnosed With Dry Eye
Brief Title: A Phase 4 Study Investigating the Efficacy of Retaine™ in Managing Signs and Symptoms Associated With Dry Eye Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ocusoft, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-110-0008
Record Dates: First submitted 2014-05-06; First posted 2014-05-15 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Dry Eye, Dry Eye Syndrome, Retaine, KCS, Keratoconjunctivitis sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

ARMS (1):
- Arm 1 (Experimental): Retain 1-2 drops, bilaterally, BID
  Interventions: Drug: Retaine™

INTERVENTIONS:
Drug: Retaine™

SUMMARY:
This study will evaluate the efficacy of Retaine™ ophthalmic emulsion in treating the signs and symptoms of dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a reported history of dry eye;
* Have a history of use or desire to use eye drops;

Exclusion Criteria:

* Have any clinically significant eye findings that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Have used Restasis® within 30 days of Visit 1;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be unwilling to submit a urine pregnancy test if of childbearing potential;
* Have a known allergy and/or sensitivity to the test article or its components;
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Tear Film Break-Up Time | Day 15
Ocular surface damage as measured by fluorescein staining | Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Andover, Massachusetts, United States